CLINICAL TRIAL: NCT05961813
Title: Evaluación de la Eficacia de Una intervención Para Dejar de Fumar en Pacientes prequirúrgicos de cirugía ortopédica o de cirugía General y urológica: Ensayo clínico Aleatorizado.
Brief Title: Intervention for Smoking Cessation in Pre-Surgical Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-483/2021
Record Dates: First submitted 2023-07-03; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Smoking; Smoking Cessation; Surgical Procedure, Unspecified
Keywords: Smoking; Smoking Cessation; Tobacco Use Disorder; Surgery
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Disorder | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Randomized, open, controlled clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group in protesic implant orthopedic surgery (Experimental): 58 patients programmed for knee or hip replacement surgeries, or spinal arthrodesis surgery who will be sent to a specialized preventive medicine consult to quit smoking.
  Interventions: Behavioral: Intensive intervention for smoking cessation
- Intervention group in general and urological surgery (Experimental): 58 patients programmed for colorrectal surgery due to colorrectal cancer, cistectomy, radical prostatectomy and partial or total nefrectomy, who will be sent to a specialized preventive medicine consult to quit smoking.
  Interventions: Behavioral: Intensive intervention for smoking cessation
- Control group in protesic implant orthopedic surgery (Active Comparator): 58 patients programmed for knee or hip replacement surgeries, or spinal arthrodesis surgery who will receive a brief intervention for smoking cessation.
  Interventions: Behavioral: Brief intervention for smoking cessation
- Control group in general and urological surgery (Active Comparator): 58 programmed for colorrectal surgery due to colorrectal cancer, cistectomy, radical prostatectomy and partial or total nefrectomy, who will receive a brief intervention for smoking cessation.
  Interventions: Behavioral: Brief intervention for smoking cessation

INTERVENTIONS:
Behavioral: Intensive intervention for smoking cessation — Patients will be given a brochure and presentation on smoking cessation and will complete 6 visits (2 before surgical intervention, 4 visits within the following 12 months), as well as follow up phone calls for progressi monitorization.
  Arms: Intervention group in general and urological surgery; Intervention group in protesic implant orthopedic surgery
Behavioral: Brief intervention for smoking cessation — Patients will be given a brochure and presentation on smoking cessation 4 weeks before surgery, as well as follow up phone calls for progressi monitorization.
  Arms: Control group in general and urological surgery; Control group in protesic implant orthopedic surgery

SUMMARY:
The goal of this clinical trial is to assess efficacy of an intensive pre-surgical intervention to quit smoking in smoking patients who will be operated on implant orthopedic surgery or general and urological surgery. The main question[s] it aims to answer are:

* Evaluate the efficacy of intensive pre surgical intervention to quit smoking compared to a brief intervention
* Evaluate the implementation of this protocol.

Participants will be randomized to 2 intervention groups (patients programmed for protesic implant orthopedic surgery in the first group, and general and urological surgery) and 2 control groups (stratified in the same manner as the intervention groups), and will be monitored through telematic check ups via phone calls.

DETAILED DESCRIPTION:
1. Subject recruitment in pre surgical anesthesiology consults, data collection and randomization within 48 hours of said visit.
2. Subjects in the intensive intervention group will be sent to a specialized Preventive Medicine consult for smoking cessation, completing 6 visits (2 before surgical intervention, 4 visits withint the following 12 months). Subjects in the control group will receive brief advice on quitting smoking through a phone call the the same day randomization is performed. Both groups will receive follow up calls at months 1, 3, 6, and 12, after surgical intervetion. All patients will have their smoking habits evaluated and the relevant data about the surgical intervention collected the day of the intervention.
3. At month 7 adecuacy of the protocol will be evaluated to assess if any modifications are necessary.
4. Data entry and quality control of the database will be performed periodically for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must 18 years old or older, and be able to consent.
* Surgery programmed for at least 4 weeks after inclusion in the study.
* Smokers

Exclusion Criteria:

* Pregnancy
* Already under treatment for smoking cessation
* Inability to consent due to cognitive impairment or language barrier.
* Non-primary knee or hip replacement surgery
* Participation in any study that forbids use of nicotine substitution therapy (dermal, oral)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Tobacco use | Evaluated at 1, 3, 6, and 12 months after surgical intervention
  Change in self reported tobacco use (smoking)

SECONDARY OUTCOMES:
Changes in concentration of exhaled CO measured with a CO-oximeter | Evaluated at recruitment, and 1, 3, 6, and 12 months after surgical intervention
  A patient will be considered as an active tobacco user if more than 6 of carboxyhemoglobin particles per million are found through the use of a CO-oximeter
Changes in rate of different type of tobbaco product users | Evaluated at recruitment, and 1, 3, 6, and 12 months after surgical intervention
  Cigarettes, cigars, rolling tobacco, etc.
Changes in tobacco use pattern | Evaluated at recruitment, and 1, 3, 6, and 12 months after surgical intervention
  Amount and frequency (daily, weekly, sporadically)
Changes in degree of nicotine dependency | Evaluated at recruitment, and 1, 3, 6, and 12 months after surgical intervention
  Fagerström test [low dependency (0-3), medium dependency (4-6), y high dependency (7-10)]
Changes in disposition to smoking cessation | Evaluated at recruitment, and 1, 3, 6, and 12 months after surgical intervention
  Prochaska and Di Clemente's model (pre contemplation, contemplation, preparation, action, maintenance or relapse)
Changes in Motivation level | Evaluated at recruitment, and 1, 3, 6, and 12 months after surgical intervention
  Richmond's test (<3 no motivation; 4-5 doubtful motivation; 6-7 moderate motivation; 8-10 high motivation)
Changes in self-efficacy | Evaluated at recruitment, and 1, 3, 6, and 12 months after surgical intervention
  Albert Bandura's social cognitive theory
Number of patients with surgical complicatoins | Hospitalization period and 90 days after surgical intervention.
  Complications will be classified as respiratory, cardiovascular, surgical wound and complications, mortality
Surgery duration | Day of intervention
  Time spent in the operation room
Need of blood transfusion | Day of intervention
  Volume of blood transfused during surgery
Hospitalization duration | Days from admitting until discharge.
  Number of days of hospitalization after surgery.
Need of new hospitalizations | 12 months after surgical intervention.
  Number of times patient is admitted to the hospital during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Eva Gavilán Castillo, RN; MSN, Principal Investigator — Vall d'Hebron Hospital
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gavilan E, Fernandez E, Minguell J, Trilla E, Sanchez JM, Espin-Basany E, Zuriguel E, Alvarez C, Montllor I, Ferre M, Aneas S, Gayubas A, Botana C, Colmenero M, Perez G, Rodriguez N, Gili N, Martinez C. Efficacy of a preoperative smoking cessation intervention in orthopedic and general and urological surgery patients: A study protocol for a randomized clinical trial. Tob Induc Dis. 2025 Oct 17;23. doi: 10.18332/tid/203550. eCollection 2025. PMID 41111564